CLINICAL TRIAL: NCT00262171
Title: Hereditary Nonpolyposis Colorectal Cancer in Taiwan-Related Genetic Study and Clinical Applications
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EC9012005
Record Dates: First submitted 2005-12-05; First posted 2005-12-06 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-03

CONDITIONS: Hereditary Nonpolyposis Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to establish the HNPCC related information in Taiwan, and to characterize relevant susceptibility genes related to colorectal cancer to provide better disease control for the high-risk people. To accomplish this objective, we will collect detailed information of the HNPCC patients and their families from the collaborative hospitals and relate the information to the risk of CRC in order to provide sound disease control system in Taiwan.

DETAILED DESCRIPTION:
HNPCC is an autosomal dominant disease that is clinically characterized by the development of colorectal cancer (CRC) at an early age (mean age 44 years old). Four genes have been known to be related to this hereditary disease. It shows an excess of synchronous and metachronous tumors as well as a preponderance of right-sided tumors (70%). Another feature has been seen among the families of the HNPCC patients is the occurrence of adenocarcinomas at other sites (particularly at the endometrial, ovary, stomach, pancreas, ureter, renal pelvis, and skin). Difficulties arise in distinguishing environmental factors and genetic predisposition for familial clustering of CRC. The discovery of HNPCC germline mutations has been momentous in that it enables a clear distinction between carriers and noncarriers for those who were previously assigned a 50% risk of germline mutation. The informed consent provided by patients is important for the process of familial study and the search for germline mutations, these will further provide information for education and counseling. HNPCC has been reported to be responsible for about 1% to 13% of all CRC. The frequency of HNPCC varies by geographical areas. The true incidence of HNPCC in Taiwan area is unclear. From year 1995 to 2000, 50 out of 4500(1.1%) patients were HNPCC according to the Amsterdam I criteria. MMR gene databases are crucial to understand the relationship between genotype and phenotype. Kindred sharing the same mutations but living in different places will provide the information to assess the contribution of environmental factors to colorectal carcinogenesis. The related clinical and basic researches are thus important for understanding the mutation spectrum of MMR genes, interaction between oncogenes, tumor suppressor genes, and roles of genetic polymorphisms in modifying MMR genes in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Select all affected individuals. If the affected is unavailable, select the spouse and adult children (20+) of these unavailable affected individuals.
* Select unaffected individuals in the following priority order:

  1. study both parents of the affected individuals;
  2. if parents are not available, study up to two siblings of each missing parent (if both parents are deceased, study four siblings - two from each parent);
  3. study up to five unaffected siblings (age 20 or older) of the affected individual; if more than five siblings are available for study, select the siblings from oldest to youngest;
  4. study up to three children (age 20 or older) of the affected individual; again, select the three oldest children if more than three are available;
  5. if the two affected individuals in the multiplex family are not siblings, (first cousins, for example, then study common grandparents - if common grandparents are not available, study siblings of these grandparents) when children of the affected individual's are studied, the child's unaffected parent will also be selected for study.

Exclusion Criteria:

* N/A

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The HNPCC patients and their families from the collaborative hospitals and relate the information to the risk of CRC in order to provide sound disease control system in Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 1014 (Actual)
Dates: Start 2002-05; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chao Hsiung, PhD., Study Director — Division of Biostatistics and Bioinformatics, National Health Research Institites; Rei-Ping Tang, PhD., Study Director — Colorectal Section, Chang Gung Memorial Hospital; Ling-Ling Hsieh, PhD., Study Director — Department of Public Health, Chang Gung University
Locations (1):
- Division of Biostatistics and Bioinformatics, National Health Research Institites, Miaoli County, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided